CLINICAL TRIAL: NCT02903693
Title: Cervical Cancer in French Guiana: Screening Between 2006-2011. Description of the Population With Invasive Cervical Cancer Between 2003-2008
Brief Title: Cervical Cancer in French Guiana: Screening Between 2006-2011
Acronym: DepCol
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: DepCol
Record Dates: First submitted 2016-09-06; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cross-Sectional Studies

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cross sectional

SUMMARY:
Given that cervical cancer is the second most frequent cancer among women in french guiana the aim of the study was to determine the screening rate among women living in French Guiana. Cervical smears are read in 2 laboratories which allowed us to compute screening rates per 100 women-years. overall the screening activity was 23.5-25.8 smears per 100 women-years. between 2006 and 2011 54% of women were screened. These baseline figures will allow to evaluate present efforts to increase the screening rate for this frequent cancer in French Guiana.

ELIGIBILITY:
Inclusion Criteria:

* women screened

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all women screened for cervical cancer using pap smear
Sampling Method: Non-Probability Sample
Enrollment: 91458 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
cervical cancer screening | 1 year (screening that year)
  Cytological examination screens for neoplasic lesion according to the Bethsda 2001, results are assessed on a yearly basis to obtain annual screening rates relative to the female population.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana, France